CLINICAL TRIAL: NCT00434564
Title: A Randomised Trial on Early Stress Nuclear Scan for Patients Presented to the Emergency Department (ED) With Chest Pain But Non-diagnostic Electrocardiography-Acute Chest Pain Treatment and Evaluation (ACTION) Study
Brief Title: Acute Chest Pain Treatment and Evaluation (ACTION) Study
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Singapore General Hospital (Other)
Collaborators: National Medical Research Council (NMRC), Singapore (Other Government); National Heart Centre Singapore (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NMRC/0517/2001
Record Dates: First submitted 2007-02-12; First posted 2007-02-13 (Estimated); Last update posted 2017-02-10 (Actual); Status verified 2017-02

CONDITIONS: Chest Pain
Keywords: Stress nuclear scan; Acute chest pain
MeSH Terms: conditions — Chest Pain

INTERVENTIONS:
Procedure: Stress nuclear scan

SUMMARY:
Objective

1. To compare the incidence of adverse cardiac events among the patients discharged after evaluation through ACTION protocol with those through conventional protocol. The adverse cardiac events for the follow-up are defined as any of the followings:

   * Cardiac related death
   * Ventricular fibrillation
   * Myocardial infarction
   * Cardiogenic shock requiring the inta-aortic balloon pump circulatory assistance
   * Acute pulmonary oedema requiring endo-tracheal intubation
2. To study the sensitivity / predictive values of the various components of ACTION :12 lead ECG ST monitoring , serial serum markers for myocardial necrosis (myoglobin, CKMB, TnT, graded exercise testing, stress tetrofosmin scan/ stress echocardiography) in predicting adverse cardiac events.

Design -prospective randomised clinical trial

Participants

-patients above 25 years of age presenting to the ED with chest pain consistent with myocardial ischaemia but with a 12 lead ECG non-diagnostic of myocardial ischaemia .

Intervention

Patients were monitored continuously with a 12 lead ECG and ST segment trend monitoring and blood will be drawn at 0,3,6 hours after arrival at ED for serial myoglobin, creatine kinase MB isoenzyme (CKMB) and Troponin T (TnT) . Patients who have ECG and blood test consistent with myocardial necrosis were admitted to the CCU. A senior doctor in the ED reviewed patients who were not admitted after 6 hours of observation.

Study Group

A stress tetrofosmin nuclear scan was done . Patients were then admitted and discharged depending on the results of the stress tetrofosmin scan.

Control group (conventional protocol)

Patients were then be admitted or discharged at the discretion of the senior ED doctor.

Measurement Patients were followed up at 1 week , 2 weeks , one month and six months for any adverse cardiac events such as cardiac related death , ventricular fibrillation , and myocardial infarction.

Statistical analysis Logistic regression analysis were used to compare the proportion of adverse events in the two treatment groups.

DETAILED DESCRIPTION:
Identifying the cause of chest pain is a challenge to the Emergency Physician.Coronary artery disease is the most common group of Emergencies that has a high potential for rapidly developing a lethal outcome.

Significant proportion of patients who presented to and released from the Emergency Department (ED)with AMI or unstable angina develop poor outcomes. This is because a large proportion of AMI present atypically.The initial single 12 lead ECG done at an ED is only 50% sensitive for AMI.Serial ECGs have been shown to improve sensitivity by 25%.Because of these limitations, physicians may admit patients with chest pain, liberally. On the other hand only 25-50 % of patients admitted to CCU without AMI are eventually determined to have Acute Coronary Syndrome.

Several serum cardiac markers such as myoglobulin, CKMB and Troponin T (TnT) are found to increase sensitivity in detecting AMI than just history and ECG. Among them TnT is a better predictor of adverse cardiac event than CKMB. Absence of TnT elevation identifies a lower risk group of patients , but not necessarily a low risk group since TnT cannot detect myocardial ischaemia in the absence of myocardial injury or myocyte cell death.

There has been some chest pain evaluation practice in the ED using the graded exercise testing to screen for severe ischaemia.

Several studies have suggested the safety of exercise testing in low risk patients presenting to ED with chest pain.The use of exercise testing has been found to be a powerful tool for prognostication.

Stress nuclear imaging was also performed at the end of 6 hours of observation instead of graded exercise stress testing alone. There will be a significant proportion of patients who will not be eligible for standard exercise treadmill stress test due to poor exercise tolerance. Even for those who underwent exercise testing, studies showed that 24.2% were inconclusive because of baseline ECG abnormalities (left ventricular hypertrophy, left bundle-branch block or patient on digoxin). Some patients may not be able to achieve the required exercise level.

Studies have shown that the mean sensitivity and specificity for graded exercise testing to detect severe coronary artery disease were 68 and 77% respectively. The sensitivity of graded exercise test for detecting single vessel disease is lower.

Stress nuclear imaging is valuable in establishing the prognosis of patients with a low likelihood of coronary artery disease. Stress nuclear scans have additive prognostic value to graded exercise test especially if the latter is abnormal or non-diagnostic.For those who cannot exercise, pharmacological stress tetrofosmin with dobutamine or adenosine will be performed instead.

The efficacy of acute chest pain evaluation centre has not been compared with a conventional protocol in a prospective randomised clinical trial.

Aims

1. To compare the incidence of adverse cardiac events among patients discharged after evaluation through ACTION with those through conventional protocol. Adverse cardiac events are defined as any of the following:

   i) Cardiac related death ii) Ventricular fibrillation iii) Myocardial infarction iv) Cardiogenic shock requiring intra-aortic balloon pump circulatory assistance v) Acute pulmonary oedema requiring endotracheal intubation
2. To study the sensitivity specificity graded exercises testing, stress tetrofosmin scan in predicting adverse cardiac event

5. Treatment Plan

First 6 hours Once informed consent was obtained, the patient was then enrolled. They were put on continuous ECG monitoring. Ten mls of blood were drawn at 0,3,6 hours after arrival at the ED for myoglobin, CKMB and TnT analysis. Blood for LDL & HDL were also drawn at 0 hour as well with the cardiac markers. The old hospital case record of patient, if available, were retrieved and previous ECG's were also compared against the new ECG.

Patients who develop recurring chest pain consistent with myocardial ischaemia, ST segment elevation or depression on continuous 12 lead ECG monitoring indicating myocardial necrosis, or have positive CKMB (> 5), Troponin T (> 0.01), were admitted to the Department of Cardiology. If the patient was not admitted at the end of 6 hours, he/she were reviewed by a ED Registrar/Associate Consultant/Consultant. The senior ED doctor reviewed the patient, his/ her 12 lead ECGs and blood results for serum markers for myocardial necrosis.

After first 6 hours - Study Group (Intervention Protocol)

The patient then underwent a stress tetrofosmin scan within 24 hours of presentation (exercise or pharmacological stress for those who cannot exercise). Tetrofosmin scans was be done at NHC or the Department of Nuclear Medicine, SGH. Patients were monitored until the test was completed. If the stress tetrofosmin scan turned out to be positive, the patient was then admitted to the hospital for further management. If the stress tetrofosmin scan was negative, the patient was released from ED with instructions for follow-up in the cardiology clinic as an outpatient.

Control Group (conventional protocol) The patient with high or intermediate risk for coronary artery disease (CAD) as defined by Agency for HealthCare Policy and Research guidelines for Unstable Angina was admitted. The indicators for coronary artery disease are definite angina, T wave inversion> 1 mm in leads with dominant R waves and diabetes. If in doubt, patients were also admitted. Patients who were discharged from the ED will be reviewed by a cardiologist at the NHC cardiac clinic within two weeks.

6. Follow Up

Patients were followed up at one month, six months and one year for any primary or secondary endpoints.

ELIGIBILITY:
Inclusion Criteria:

* 25 years and above
* Chest pain suggestive of the angina
* 12 leads ECG non-diagnostic for myocardial ischaemia or AMI
* diabetes mellitus
* family history of young AMI (less than 50 years old) There is no lower limit of age for those patients in the last two categories

Exclusion Criteria:

* ECG diagnostic of AMI or acute myocardial ischaemia (as defined by the new Q wave , ST elevation or depression greater than 1mm or 0.1 millivolts in two or more contiguous leads)
* Congestive heart failure or hypotensive patients
* Persistent chest pain consistent with unstable angina

Min Age: 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1690
Dates: Start 2000-08; Study Completion 2002-05

PRIMARY OUTCOMES:
Cardiac related death
Ventricular Fibrillation
Myocardial Infarction
Cardiogenic shock requiring intra-aortic balloon pump circulatory assistance
Acute pulmonary oedema requiring endotracheal intubation

SECONDARY OUTCOMES:
Requirement of emergency coronary revascularisation procedures like Percutaneous Transluminal Coronary Angioplasty (PTCA) or Coronary Artery Bypass Graft (CABG)

CONTACTS AND LOCATIONS:
Overall Officials: Lim S Han, MBBS, FRCS, Principal Investigator — Department of Emergency Medicine, Singapore General Hospital
Locations (1):
- Singapore General Hospital, Singapore, Singapore

REFERENCES:
- [Background] Lee TH, Rouan GW, Weisberg MC, Brand DA, Acampora D, Stasiulewicz C, Walshon J, Terranova G, Gottlieb L, Goldstein-Wayne B, et al. Clinical characteristics and natural history of patients with acute myocardial infarction sent home from the emergency room. Am J Cardiol. 1987 Aug 1;60(4):219-24. doi: 10.1016/0002-9149(87)90217-7. PMID 3618483
- [Background] McCarthy BD, Beshansky JR, D'Agostino RB, Selker HP. Missed diagnoses of acute myocardial infarction in the emergency department: results from a multicenter study. Ann Emerg Med. 1993 Mar;22(3):579-82. doi: 10.1016/s0196-0644(05)81945-6. PMID 8442548
- [Background] Pozen MW, D'Agostino RB, Selker HP, Sytkowski PA, Hood WB Jr. A predictive instrument to improve coronary-care-unit admission practices in acute ischemic heart disease. A prospective multicenter clinical trial. N Engl J Med. 1984 May 17;310(20):1273-8. doi: 10.1056/NEJM198405173102001. PMID 6371525
- [Background] Kannel WB, Abbott RD. Incidence and prognosis of unrecognized myocardial infarction. An update on the Framingham study. N Engl J Med. 1984 Nov 1;311(18):1144-7. doi: 10.1056/NEJM198411013111802. PMID 6482932
- [Background] Gibler WB, Runyon JP, Levy RC, Sayre MR, Kacich R, Hattemer CR, Hamilton C, Gerlach JW, Walsh RA. A rapid diagnostic and treatment center for patients with chest pain in the emergency department. Ann Emerg Med. 1995 Jan;25(1):1-8. doi: 10.1016/s0196-0644(95)70347-0. PMID 7802357
- [Background] McGuinness JB, Begg TB, Semple T. First electrocardiogram in recent myocardial infarction. Br Med J. 1976 Aug 21;2(6033):449-51. doi: 10.1136/bmj.2.6033.449. PMID 953603
- [Background] Behar S, Schor S, Kariv I, Barell V, Modan B. Evaluation of electrocardiogram in emergency room as a decision-making tool. Chest. 1977 Apr;71(4):486-91. doi: 10.1378/chest.71.4.486. PMID 856546
- [Background] Gibler WB, Gibler CD, Weinshenker E, Abbottsmith C, Hedges JR, Barsan WG, Sperling M, Chen IW, Embry S, Kereiakes D. Myoglobin as an early indicator of acute myocardial infarction. Ann Emerg Med. 1987 Aug;16(8):851-6. doi: 10.1016/s0196-0644(87)80521-8. PMID 3619163
- [Background] Gibler WB, Lewis LM, Erb RE, Makens PK, Kaplan BC, Vaughn RH, Biagini AV, Blanton JD, Campbell WB. Early detection of acute myocardial infarction in patients presenting with chest pain and nondiagnostic ECGs: serial CK-MB sampling in the emergency department. Ann Emerg Med. 1990 Dec;19(12):1359-66. doi: 10.1016/s0196-0644(05)82598-3. PMID 2240745
- [Background] Katus HA, Remppis A, Neumann FJ, Scheffold T, Diederich KW, Vinar G, Noe A, Matern G, Kuebler W. Diagnostic efficiency of troponin T measurements in acute myocardial infarction. Circulation. 1991 Mar;83(3):902-12. doi: 10.1161/01.cir.83.3.902. PMID 1999039
- [Background] Gianrossi R, Detrano R, Mulvihill D, Lehmann K, Dubach P, Colombo A, McArthur D, Froelicher V. Exercise-induced ST depression in the diagnosis of coronary artery disease. A meta-analysis. Circulation. 1989 Jul;80(1):87-98. doi: 10.1161/01.cir.80.1.87. PMID 2661056
- [Background] Sawada SG, Ryan T, Conley MJ, Corya BC, Feigenbaum H, Armstrong WF. Prognostic value of a normal exercise echocardiogram. Am Heart J. 1990 Jul;120(1):49-55. doi: 10.1016/0002-8703(90)90159-u. PMID 2360517
- [Background] Braunwald E, Jones RH, Mark DB, Brown J, Brown L, Cheitlin MD, Concannon CA, Cowan M, Edwards C, Fuster V, et al. Diagnosing and managing unstable angina. Agency for Health Care Policy and Research. Circulation. 1994 Jul;90(1):613-22. doi: 10.1161/01.cir.90.1.613. PMID 8026048